CLINICAL TRIAL: NCT04767711
Title: Prevention of Glucocorticoid Induced Impairment of Bone Metabolism - A Randomized, Placebo-Controlled, Single Centre Clinical Trial
Brief Title: Prevention of Glucocorticoid Induced Impairment of Bone Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Mattias Lorentzon, Professor, Chief Physician, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCreuteri
Record Dates: First submitted 2021-02-12; First posted 2021-02-23 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L. reuteri (Active Comparator): Capsules of freeze-dried L. reuteri 6475 of 5x10E9 colony-forming units (CFU) mixed with maltodextrin powder and 200 IU of cholecalciferol, taken twice daily for 30 days, yielding a total daily dose of 1x10E10 L.reuteri CFU and 400 IU of cholecalciferol per day. Oral glucocorticoid 25 mg daily for 7 days.
  Interventions: Dietary Supplement: Lactobacillus reuteri ATCC PTA 6475 (L. reuteri 6475); Drug: Prednisolone
- Placebo (Placebo Comparator): Placebo product identical to the active product (L. reuteri) in taste and appearance but without the active component, orally twice daily, for 30 days.The placebo product contains 200 IU cholecalciferol per dose, yielding a total dose of cholecalciferol of 400 IU per day. Oral glucocorticoid 25 mg daily for 7 days.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri ATCC PTA 6475 (L. reuteri 6475) — L.reuteri with cholecalciferol compared to cholecalciferol only.
  Arms: L. reuteri
Drug: Prednisolone — Oral glucocorticoid 25 mg daily for 7 days.

SUMMARY:
Glucocorticoid (GC) therapy is used to treat a variety of inflammatory conditions such as rheumatoid arthritis, inflammatory bowel disease, bronchial asthma, allergies, ankylosing spondylitis and some forms of cancers. Despite the well-known side-effects, GC treatment is widely used. Oral GC therapy leads to a rapid and profound effects on bone metabolism, with increased osteoblast apoptosis and prolonged osteoclast survival, which increases bone resorption, resulting in bone loss, and a subsequent increased fracture risk. Within days of high dose oral GC, glucose tolerance decreases and bone turnover is shifted in favour of less bone formation and increased bone resorption. Bone formation and bone resorption can be estimated by measuring serum bone turnover markers.

The gut microbiota is involved in regulating bone metabolism and recently it was demonstrated that Lactobacillus reuteri 6475 (LR) could reduce bone loss over 12 months by half in older women. In a recent experimental study, it was discovered that mice treated either with broad spectrum antibiotics, eradicating gut microbiota, or with LR did not experience GC induced bone loss in the spine and femur. L. reuteri has been widely studied in clinical trials and has been shown to have probiotic, health-promoting effects in both adults and children.

The aim of this planned randomized, double-blind, placebo-controlled trial is to investigate if daily supplementation with LR, compared to placebo, can prevent the negative effects of oral glucocorticoid (GC) on bone turnover and on blood glucose regulation in healthy young adult men and women.

If LR is able to prevent deleterious side effects, such as bone loss and impaired glucose tolerance, of oral GC treatment, the probiotic could potentially be recommended and used to improve health in a substantial yearly number of patients treated with GC.

DETAILED DESCRIPTION:
By advertising in newspapers, in shops, health clubs, in public places, and on social media platforms, and by contacting interested persons (by mail and phone) identified publicly available websites (e.g. www.ratsit.se), 46 young, healthy men and women will be recruited, to participate in the study. Study subjects will be contacted by phone and receive more information regarding the study and undergo a preliminary evaluation about eligibility to participate. Detailed study information will be sent by mail to study subjects. At the screening visit, participants will receive information about the study verbally, and if participants sign the informed consent form, participants will undergo a test of fasting blood glucose, HbA1c, and an oral glucose tolerance test (OGTT). A standardized self-reported questionnaire will be used to collect information at the screening visit about smoking habits, calcium intake, medical history, medications, previous fractures, physical activity, and diet habits. Eligible participants are then invited to the randomization visit. At the randomization visit, the study subjects will be asked to refrain from physical exercise, other than walking and keep an unchanged normal diet from study day 14. Randomization will be carried out by the supplier of LR (BioGaiaAB). The investigators will not have access to the randomization code and blinding will be maintained until study end and database lock. After randomization, study participants will consume either LR or placebo for 30 days. After the 14-day run-in period, all participants will start taking 25 mg of oral prednisolone every morning for 7 days. At the 14-day visit, a 24-hour glucose monitoring for the following 10 days will be started. At the next visit on day 16, fasting blood samples will be drawn in the morning (7-9 am), feces samples provided (within 24 hours of collection) and participants will start the oral GC treatment on that visit after blood samples have been drawn. At the 19-, 23- and 30-day visits, blood samples will be drawn in the morning (7-9 am for all visits, prior to taking the GC dose). Feces samples will also be collected at these visits. Included participants will be asked to come to the clinic and report compliance and possible adverse events during the duration of the study and at all visits.

Analyses.

Questionnaires:

A standardized questionnaire will be used to collect information at the screening visit about smoking habits, calcium intake, medical history (e.g. stroke, rheumatoid arthritis, and diabetes), medications, and previous fractures. Current physical activity and diet habits will be assessed by self-reported questionnaires (IPAQ and FFQ) at baseline. Daily intake of calcium will be calculated from the questionnaires about calcium-containing foods (e.g. dairy products, vegetables etc). Gastrointestinal symptoms will be analyzed using the GSRS questionnaire.

Serum, plasma, and stool analyses:

Serum and plasma will be collected in the morning (fasting), frozen, and stored at -80° C until further analyses. Samples from day 16 will be drawn prior to oral GC treatment start. A maximum of 30 ml of blood will be collected at each visit. Fasting blood glucose will be analyzed using fresh blood at screening (with the addition of HbA1c at screening), and days 16 (GC start), 19, 23, and 30. Serum and plasma samples will be frozen immediately and kept until analysis. Analyses of serum or plasma and bone markers (osteocalcin, P1NP, and CTX) will be performed using commercially available immunosorbent assays. Stool samples will be collected within 24 hours since produced and stored at -80oC until further analysis.

Oral glucose tolerance test (OGTT):

At the screening visit, a morning fasting blood glucose will be measured, followed by ingestion of 24 cl of glucose syrup, containing 75 grams of sugar. After 2 hours another blood glucose measurement will be performed. Inclusion in the study will depend on having a normal fasting blood glucose (≤6 mmol/l) and OGTT (<7.8 mmol/l).

Markers of intestinal permeability and intestinal inflammation:

Analyses of markers for intestinal permeability (endotoxin analysis, PyroGeneTM Recombinant Factor C Endpoint Fluorescent Assay) will be performed using a fluorescent assay at day 16, day 19, and day 23. Markers of intestinal inflammation (lipocalin-2 and calprotectin) will also be analyzed in feces and serum.

Analyses of gut microbiota - exploratory analyses:

DNA from feces samples will be isolated using a well-validated protocol and perform PCR to amplify the variable regions (V4) of the bacterial 16S rRNA gene using barcoded primers. Metagenome analyses of all samples will also be performed.

Continuous glucose monitoring:

On study day 14, continuous glucose monitoring (CGM) will be started, allowing a 48-hour observation period prior to commencement of oral prednisolone dosing. CGM will be used from day 14 until prednisolone treatment cessation on day 23. The Dexcom G6 system will be used for CGM on all participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, 18-45 years old.
* Stated availability throughout the entire study period.
* Ability to understand study instructions and willingness to adhere to the protocol.
* Signed informed consent.
* Vaccinated for Covid-19

Exclusion Criteria:

* History of diabetes or glucose intolerance, defined as an abnormal oral glucose tolerance test (OGTT).
* Obesity, BMI>30 kg/m2
* History of adrenal disease or impairment.
* Previous (within the last 5 years) or current use of antiresorptive therapy, including systemic hormone therapy (estrogen), bisphosphonates, strontium ranelate or denosumab.
* Participation in other clinical trials.
* Current antibiotics treatment or within the last 2 months prior to inclusion.
* Current and within the past 2 months use of probiotic supplement.
* Untreated hyperthyroidism or hyperthyroidism within the last 5 years.
* Known untreated hyperparathyroidism.
* Rheumatoid arthritis.
* Diagnosed with disease causing secondary osteoporosis, including chronic obstructive pulmonary disease, inflammatory bowel disease, celiac disease, or diabetes mellitus.
* Recently diagnosed malignancy (within the last 5 years).
* Systemic skeletal disease (including e.g. Paget's disease and osteogenesis imperfecta).
* Any systemic disease that could affect bone loss, as judged by the investigator.
* Oral corticosteroid use.
* History of peptic ulcer.
* Diagnosed osteoporosis.
* Current smoking or other use of nicotine containing products.
* Pregnancy.
* History of any psychiatric disorder, including psychosis, depression, anxiety disorder and bipolar disorder.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Change in bone turnover marker serum osteocalcin | Baseline (day 16) to day 23
  Between group percent change in bone turnover markers osteocalcin between baseline (day 16, prior to GC treatment start) and day 23 (7 days after starting oral GC).
Change in bone turnover marker serum PINP | Baseline (day 16) to day 23
  Between group percent change in bone turnover markers serum PINP between baseline (day 16, prior to GC treatment start) and day 23 (7 days after starting oral GC).
Change in bone turnover marker serum CTX | Baseline (day 16) to day 23
  Between group per cent change in bone turnover marker serum CTX between baseline (day 16, prior to GC treatment start) and day 23 (7 days after starting oral GC).

SECONDARY OUTCOMES:
Change in blood glucose levels | Day 14-16 to day 16-23
  Change in blood glucose levels (area under the curve, mmol/L) using continuous glucose monitoring (CGM) between baseline (day 14-16) and days 16-23.
Change in serum marker of intestinal permeability - endotoxin levels | Baseline (day 16) to day 23
  Change between baseline (day 16) and day 23 in serum markers of intestinal permeability (endotoxin levels, % change).
Change in feces marker lipocalin-2 of intestinal inflammation | Baseline (day 16) and day 23
  Percent change between baseline (day 16) and day 23 in feces marker lipocalin-2 of intestinal inflammation.
Change in feces marker calprotectin of intestinal inflammation | Baseline (day 16) and day 23
  Percent change between baseline (day 16) and day 23 in feces marker calprotectin of intestinal inflammation.
Change in serum marker lipocalin-2 of intestinal inflammation | Baseline (day 16) and day 23
  Percent change between baseline (day 16) and day 23 in serum marker lipocalin-2 of intestinal inflammation
Change in serum marker calprotectin of intestinal inflammation | Baseline (day 16) and day 23
  Percent change between baseline (day 16) and day 23 in serum marker calprotectin of intestinal inflammation.
Change in the gut microbiota composition | Baseline (day 16) and day 23
  Change in the gut microbiota composition between baseline (day 16) and day 23.

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Lorentzon, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Geriatric Medicine, Sahlgrenska University Hospital, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nilsson AG, Sundh D, Backhed F, Lorentzon M. Lactobacillus reuteri reduces bone loss in older women with low bone mineral density: a randomized, placebo-controlled, double-blind, clinical trial. J Intern Med. 2018 Sep;284(3):307-317. doi: 10.1111/joim.12805. Epub 2018 Jul 22. PMID 29926979
- [Derived] Gregori G, Johansson L, Silberberg L, Imberg H, Magnusson P, Lind M, Lorentzon M. Prevention of glucocorticoid-induced impairment of bone metabolism-a randomized, placebo-controlled, single centre proof-of-concept clinical trial. JBMR Plus. 2025 Feb 17;9(4):ziaf031. doi: 10.1093/jbmrpl/ziaf031. eCollection 2025 Apr. PMID 40162303